CLINICAL TRIAL: NCT06083896
Title: Minimally-invasive Stabilization of Pelvic Metastases With Photodynamic Nails: A Multi-center Prospective Study of Functional Outcome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0292; NCI-2023-08747 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Photodynamic nails — stab incision is made at the entry site

SUMMARY:
Determine whether patients exhibit early functional improvement after minimally-invasive placement of Illuminoss photodynamic nails for peri-acetabular pelvic metastasis at 3 months following procedure

DETAILED DESCRIPTION:
Primary Objectives

1. Evaluate whether patients exhibit early functional improvement after minimally-invasive placement of Illuminoss photodynamic nails for peri-acetabular pelvic metastasis at 3 months following procedure

Secondary Objectives

1. Evaluate whether the procedure relieves pain
2. Evaluate radiographic stability of the implant
3. Evaluate functional outcome at earlier time points (2 weeks or 6 weeks) and at 6 months and possibly later time points
4. Evaluate reoperation rate and complications

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed malignancy from prior biopsy of the primary tumor or a metastatic site. Patients with carcinoma, myeloma, and lymphoma may be included in the study. Patients should have metastatic involvement of the periacetabular region that is visible radiographically. Biopsy of acetabular disease is not required for this study.
* Age ≥18 years (Illuminoss is approved only for skeletally mature patients)
* Suitable candidate for general anesthesia
* Ability to understand and the willingness to sign a written informed consent document.
* Able and willing to fill out pre-operative and post-operative functional outcome surveys
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 50,000/mcL

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness (e.g., recent pneumonia or myocardial infarction that would significantly increase risk of general anesthesia)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the risk of general anesthesia and radiation exposure (fluoroscopy) to the fetus
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dental resins or PET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion, up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org